CLINICAL TRIAL: NCT05642078
Title: A Randomized, Blind, Position-controlled Phase III Clinical Trial to Evaluate the Immunogenicity and Safety of Quadrivalent Influenza Virus Split Vaccine in 6-35 Months of Age
Brief Title: Phase Ⅲ Clinical Study of Quadrivalent Influenza Virus Split Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LKM-2022-FIn001
Record Dates: First submitted 2022-11-25; First posted 2022-12-08 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-10

CONDITIONS: Prevention of Influenza

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational Vaccine(Low dose group) (Experimental): Quadrivalent influenza vaccine(Split Virion),Inactivated，Produced by Anhui Zhifei Longcom Biopharmceutical Co., Ltd.；0.25mL/branch, each contains 7.5 μg H1N1, H3N2, B(V), B(Y) hemagglutinin.Subjects were vaccinated with one dose of vaccine on day 0 and day 28 respectively.
  Interventions: Biological: Investigational Vaccine(0.25ml/vial)
- Investigational Vaccine(High dose group) (Experimental): Quadrivalent influenza vaccine(Split Virion),Inactivated，Produced by Anhui Zhifei Longcom Biopharmceutical Co., Ltd.；0.5mL/branch, each contains 15 μg H1N1, H3N2, B(V), B(Y) hemagglutinin.Subjects were vaccinated with one dose of vaccine on day 0 and day 28 respectively.
  Interventions: Biological: Investigational Vaccine(0.5ml/vial)
- Active compared Vaccine (Active Comparator): Influenza Vaccine(Split Virion),Inactivated Quadrivalent,Produced by Hualan Biological Vaccine Co., Ltd.;0.25mL/branch,each contains 7.5 μg H1N1, H3N2, B(V), B(Y) hemagglutinin.Subjects were vaccinated with one dose of vaccine on day 0 and day 28 respectively.
  Interventions: Biological: Active compared Vaccine

INTERVENTIONS:
Biological: Investigational Vaccine(0.25ml/vial) — Subjects were vaccinated with a dose of low-dose Investigational vaccine on day 0 and day 28 respectively.The site of inoculation for infants aged 6-11 months is the anterolateral thigh, and the site of inoculation for infants aged 12-35 months is the lateral deltoid muscle of the upper arm.
  Arms: Investigational Vaccine(Low dose group)
Biological: Investigational Vaccine(0.5ml/vial) — Subjects were vaccinated with a dose of high-dose Investigational vaccine on day 0 and day 28 respectively.The site of inoculation for infants aged 6-11 months is the anterolateral thigh, and the site of inoculation for infants aged 12-35 months is the lateral deltoid muscle of the upper arm.
  Arms: Investigational Vaccine(High dose group)
Biological: Active compared Vaccine — Subjects were vaccinated with a dose of active compared vaccine on day 0 and day 28 respectively.The site of inoculation for infants aged 6-11 months is the anterolateral thigh, and the site of inoculation for infants aged 12-35 months is the lateral deltoid muscle of the upper arm.
  Arms: Active compared Vaccine

SUMMARY:
A randomized, blind, positive vaccine control trial was designed.A total of 2550 subjects aged 6-35 months were randomly assigned to the low dose (0.25ml/ dose) group, the high dose (0.5ml/ dose) group and the control group in a ratio of 1:1:1. They were inoculated with 2 doses of quadrivalent influenza virus split vaccine (experimental vaccine or control vaccine) at 0 and 28 days of immunization program to observe the Immunogenicity and safety.

DETAILED DESCRIPTION:
A randomized, blind, positive vaccine control trial was designed.A total of 2550 subjects aged 6-35 months were randomly assigned to the low dose (0.25ml/ dose) group, the high dose (0.5ml/ dose) group and the control group in a ratio of 1:1:1. They were inoculated with 2 doses of quadrivalent influenza virus split vaccine (experimental vaccine or control vaccine) at 0 and 28 days of immunization program to observe the Immunogenicity and safety.

Immunogenicity observation Venous blood (2.5-3.0ml) was collected from all subjects before the first dose and 30 days after the full dose, and serum was separated for detection of Hemagglutination Inhibition antibodies against four influenza virus serotypes (H1N1, H3N2, B (V), B (Y)).

Safety observation All AE within 30 minutes of each dose, solicited adverse events at 0-7 days, non-solicited adverse events at 0-28 days (first dose) /30 days (second dose), and all serious adverse events from the first dose to 6 months after the full dose were collected.

ELIGIBILITY:
Inclusion Criteria:

* （1）The age at the time of joining the group is 6-35 months old, and can provide legal identification.
* （2）The legal guardian of the subject voluntarily agreed to the child's participation in the study and signed the informed consent form.
* （3）The legal guardian of the subject has the ability to understand the research procedures and to participate in the follow-up of all plans.
* （4）On the day of joining the group, the armpit temperature was less than 37.3 ℃.

Exclusion Criteria:

* （1）Before joining the group, they have been vaccinated against influenza in this epidemic season or have plans to receive influenza vaccination during the study period.
* （2）Suffered from influenza disease in the past 3 months (confirmed by clinical, serological or microbiological methods)
* （3）Babies (6-11 months old) are born with a gestational age of < 37 weeks or ≥ 42 weeks.
* （4）Babies (6-11 months old) weigh less than 2.5kg or > 4.0kg at birth and are not suitable to participate in this study.
* （5）Babies (6-11 months old) are born during abnormal labor (dystocia, instrumental delivery, excluding caesarean section) or have a history of asphyxia or neurological damage
* （6）Previous history of severe allergy to any vaccine / drug or to any component of the test vaccine (including ovalbumin, etc.), such as anaphylactic shock, anaphylactic laryngeal edema, anaphylactoid purpura, thrombocytopenic purpura, local allergic necrotic reaction (Arthus reaction), severe urticaria, etc.
* （7）Have a history of severe allergy to eggs or egg proteins, such as angioneurotic edema, dyspnea, chest tightness, or repeated vomiting due to eating eggs, or even use epinephrine or other emergency medical treatment, especially those who develop symptoms within a short period of time (minutes to hours) after eating.
* （8）Acute disease or acute attack of chronic disease occurred within 3 days before vaccination.
* （9）Before entering the group, the interval between other live vaccines was less than 7 days, and the interval between live attenuated vaccines was less than 14 days.
* （10）Use antipyretic analgesic or antiallergic drugs within 3 days before entering the group.
* （11）Have used other research or unregistered products (drugs or vaccines) within 1 month before joining the group, or plan to participate in other clinical studies after joining the group.
* （12）Long-term use of immunosuppressants or other immunomodulatory drugs within the first 3 months (defined as continuous use for more than 14 days), such as glucocorticoid dose ≥ 0.5mg/kg/ days (inhaled and topical glucocorticoids are not restricted)
* （13）Received blood or blood-related products within 6 months before joining the group (hepatitis B immunoglobulin acceptable).
* （14）Has been diagnosed with congenital or acquired immunodeficiency disease.
* （15）Suffering from serious diseases or congenital malformations that may interfere with the conduct or completion of research (including, but not limited to, respiratory diseases such as asthma or chronic bronchitis, Down syndrome, thalassemia, heart disease, nephropathy, autoimmune diseases, Guillain-Barre syndrome, severe developmental disorders, severe eczema, etc.)
* （16）Has been diagnosed with systemic diseases that may interfere with the conduct or completion of research, such as tuberculosis, viral hepatitis and / or human immunodeficiency virus HIV infection.
* （17）Have a history of convulsions, epilepsy, encephalopathy and mental illness or family history.
* （18）There are contraindications for intramuscular injection, such as having been diagnosed with thrombocytopenia, any coagulation disorder or receiving anticoagulant treatment.
* （19）No spleen, functional no spleen, and no spleen or splenectomy caused by any condition.
* （20）Plan to move out of Hong Kong before the end of the study or for a long period of time during the visit to the project study.
* （21）The researchers believe that the subjects have any situation that may interfere with the evaluation of the purpose of the study.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2550 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Immunogenicity end point 1 | 30 days after the whole vaccination
  30 days after the whole vaccination, the seroconversion rate of serum Hemagglutination Inhibition antibodies of influenza viruses H1N1, H3N2, B(V) and B(Y) were observed.
Immunogenicity end point 2 | 30 days after the whole vaccination
  30 days after the whole vaccination, the geometric mean titer of serum Hemagglutination Inhibition antibodies of influenza viruses H1N1, H3N2, B(V) and B(Y) were observed.
Immunogenicity end point 3 | 30 days after the whole vaccination
  30 days after the whole vaccination, the seroprotection rate of serum Hemagglutination Inhibition antibodies of influenza viruses H1N1, H3N2, B(V) and B(Y) were observed.
Immunogenicity end point 4 | 30 days after the whole vaccination
  30 days after the whole vaccination, the geometric mean increase of serum Hemagglutination Inhibition antibodies of influenza viruses H1N1, H3N2, B(V) and B(Y) were observed.
Safety end point 1 | Within 30 days from the first dose to the whole course of vaccination
  Incidence and severity distribution of all adverse events within 30 days from the first dose to the whole course of vaccination.
Safety end point 2 | Within 30 minutes after each dose
  Incidence and severity distribution of total AE within 30 minutes after each dose.
Safety end point 3 | Within 7 days after each dose
  Incidence and severity distribution of conscriptive adverse events within 7 days after each dose.
Safety end point 4 | Within 0-28 days after first dose vaccination and 0-30 days after second dose vaccination
  Incidence and severity distribution of non-aggregative adverse events within 0-28 days after first dose vaccination and 0-30 days after second dose vaccination.
Safety end point 5 | Within 6 months from the first dose to the whole course of vaccination
  Incidence of serious adverse events within 6 months from the first dose to the whole course of vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Huang, Bachelor, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China